CLINICAL TRIAL: NCT03163329
Title: A Prospective, Randomized, Controlled, Multi-Center Study to Establish the Safety and Effectiveness of Transcatheter Aortic Valve Raplacemet in Intermediate Risk Patients Who Have Severe, Calcific, Bicuspid, Aortic Stenosis Requiring Aortic Valve Replacement
Brief Title: The Safety and Effectiveness of Transcatheter Aortic Valve Raplacemet in Intermediate Risk Patients With Bicuspid Aortic Stenosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Yongjian Wu, Clinical Professor, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AS-20170520
Record Dates: First submitted 2017-05-20; First posted 2017-05-23 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAVR group (Experimental)
  Interventions: Procedure: TAVR
- SAVR group (Active Comparator)
  Interventions: Procedure: SAVR

INTERVENTIONS:
Procedure: TAVR — Transcatheter Aortic Valve Replacement
  Arms: TAVR group
Procedure: SAVR — Surgical Aortic Valve Replacement
  Arms: SAVR group

SUMMARY:
Previous trials have shown that TAVR was a noninferior alternative to surgery in patients with severe aortic stenosis at intermediate surgical risk. However, patients with congenital bicuspid valve have been excluded in those trials. The purpose of this trial is to determine the safety and effectiveness of TAVR in intermediate-risk patients with bicuspid aortic valve stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Severe, calcific bicuspid aortic stenosis.
2. Heart team agrees the patient has a risk of operative mortality and has an STS <8 and >3.
3. The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.

Exclusion Criteria:

1. Ilio-femoral vessel characteristics that would preclude safe placement of the introducer sheath.
2. Evidence of an acute myocardial infarction ≤ 1 month (30 days) before randomization.
3. Severe aortic regurgitation (>3+).
4. Severe mitral regurgitation (>3+).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality, all stroke, and re-hospitalization | 1 year post procedure
  This composite endpoint will be evaluated as a non-inferiority analysis based on a relative non-inferiority margin of 35%